CLINICAL TRIAL: NCT06797557
Title: Biochemical, 2D and 3D Ultrasonographic Predictors of Pregnancy Outcome in Women With Threatened Abortion: A Prospective Cohort Study
Brief Title: Biochemical, 2D and 3D Ultrasonographic Predictors of Pregnancy Outcome in Women With Threatened Abortion
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Other Study IDs: N 363
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Threatened Miscarriage
MeSH Terms: conditions — Abortion, Threatened

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 ml venous blood samples were collected for hormonal measurement from the brachial vein of the patients in plain tubes. All blood samples were centrifuged for 10 minutes at 1,000 RPM at room temperature and the serum extracted and frozen at -20oC.
  * Serum HCG concentrations (intact HCG plus the HCG β-subunit) were quantified using an automated immunoassay technique and expressed in IU/L using the World Health Organization Third International Reference.
  * Progesterone assay principle combines an enzyme immunoassay competition method with final fluorescent detection. Levels were quantified using an automated immunoassay and expressed in ng/mL
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 2D Ultrasound — * Crow- rump length (CRL) measurement using 2D ultrasound. Proper measurement of the CRL was done according to obtaining a true, unflexed, longitudinal section of the embryo or fetus, with the end-points of the crown (the top of the head) and rump (the end of the trunk) clearly defined, and then placing the calipers correctly on these defined end-points.
  * Yolk sac diameter (largest outer to outer measure).
  * Mean gestational sac diameter (arithmetic mean of 3 diameters).
  * Embryonic heart rate. the heart rate was determined from M-mode tracings using electronic calipers .The sweep speed was set at 4 s and the calculation of the heart rate was made by measuring the time interval of two cardiac cycles, using clearly identified points in the M-mode tracing
Diagnostic Test: 3D ultrasound — 3D ultrasound rotational VOCAL method was used. YSV measurement (axial, sagittal and coronal). The sagittal plane was chosen as the reference plane and 'scanned' to obtain the longest axis of the yolk sac. Then a magnification of image was used and the yolk sac moved to the center of the plane. The VOCAL switch was then activated using a 30° rotation angle and the manual setting. Calipers were positioned on the superior and inferior extremities of the structure and after obtaining six sequential planes, the equipment automatically displayed the yolk sac as a 3D image with its volume in cm3

SUMMARY:
Three or two measurements (according to GA) using 2D and 3D ultrasound examinations will be done at initial assessment of the participants then after 1 to 2 weeks and at the end of the 12th week of gestation

DETAILED DESCRIPTION:
First ultrasound scans: between 6 and 11 weeks of gestation that included the following:

* Crow- rump length (CRL) measurement using 2D ultrasound. Proper measurement of the CRL was done according to obtaining a true, unflexed, longitudinal section of the embryo or fetus, with the end-points of the crown (the top of the head) and rump (the end of the trunk) clearly defined, and then placing the calipers correctly on these defined end-points.
* Yolk sac diameter (largest outer to outer measure).
* Mean gestational sac diameter (arithmetic mean of 3 diameters).
* Embryonic heart rate. the heart rate was determined from M-mode tracings using electronic calipers .The sweep speed was set at 4 s and the calculation of the heart rate was made by measuring the time interval of two cardiac cycles, using clearly identified points in the M-mode tracing
* For volume calculation, 3D ultrasound rotational VOCAL method was used. YSV measurement (axial, sagittal and coronal). The sagittal plane was chosen as the reference plane and 'scanned' to obtain the longest axis of the yolk sac. Then a magnification of image was used and the yolk sac moved to the center of the plane. The VOCAL switch was then activated using a 30° rotation angle and the manual setting. Calipers were positioned on the superior and inferior extremities of the structure and after obtaining six sequential planes, the equipment automatically displayed the yolk sac as a 3D image with its volume in cm3.

Follow up scans was done one to two weeks later according the patient condition then at the end of 1st trimester where the previously mentioned parameters were measured.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 -39 years
* BMI 18-25 kg/m2
* Singleton pregnancy between 6 to 11 gestational weeks of pregnancy.
* First trimester threatened abortion is usually diagnosed in women with history of vaginal bleeding or spotting and/or abdominal pain in whom a live embryo can visualized on scan
* Gestational age (GA) calculated by the last menstrual period date (LMP) in women with sure dates and regular menstrual cycles and confirmed by transvaginal sonography performed up to the 11th gestational week, using the crown-rump length

Exclusion Criteria:

* Uterine malformations or pathology as submucous myoma
* Cervical abnormalities as polypi or severe chronic cervicitis
* Chronic medical conditions as uncontrolled diabetes or hypertension
* Smoking or drug abuse during this pregnancy
* Pregnancies resulting from infertility treatments and assisted reproductive techniques.
* Women with exogenous progesterone support
* Use of abortion induction drugs\
* First trimester vaginal bleeding or spotting and/or abdominal pain and diagnosed by ultrasound as missed (absence of cardiac activity within fetal pole), incomplete (endometrial thickness between 5 to 15 mm), complete (thin and regular endometrium), anembryonic (gestational sac without a detectable fetal pole) and ectopic (+ve pregnancy test with empty gestational sac

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women with threatened abortion
Study Population: One hundred and twenty women with threatened abortion.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks of gestational age
  continuation of pregnancy beyond 12 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided